CLINICAL TRIAL: NCT00528866
Title: Adjuvant 3DCRT/IMRT in Combination With Androgen Suppression and Docetaxel for High Risk Prostate Cancer Patients Post-Prostatectomy: A Phase II Trial
Brief Title: Radiation Therapy, Androgen Suppression, and Docetaxel in Treating Patients With High-Risk Prostate Cancer Who Have Undergone Radical Prostatectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-0621; CDR0000563917; NCI-2009-00740 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2007-09-10; First posted 2007-09-12 (Estimated); Results first posted 2017-06-06 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2018-05

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — bicalutamide; Docetaxel; Flutamide; Gonadotropin-Releasing Hormone; Radiotherapy, Conformal; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Androgen suppression + RT + docetaxel (Experimental): LHRH agonist and oral antiandrogen (flutamide or bicalutamide), radiation therapy (RT), and docetaxel
  Interventions: Drug: bicalutamide; Drug: docetaxel; Drug: flutamide; Drug: LHRH agonist; Radiation: 3-dimensional conformal radiation therapy; Radiation: radiation therapy

INTERVENTIONS:
Drug: bicalutamide — 50 mg (one tablet) daily orally for 6 months, starting within 6 months after registration
Drug: docetaxel — 75 mg/m2 IV over 1 hour on day 1 of each cycle q21 days for 6 cycles, starting 3-6 weeks after completion of radiation therapy
Drug: flutamide — 250 mg (two 125-mg capsules) three times daily (total 750 mg) orally for 6 months, starting within 6 months after registration
Drug: LHRH agonist — LHRH agonist (such as leuprolide, goserelin, buserelin, or triptorelin) for 6 months, starting within 6 weeks after registration
Radiation: 3-dimensional conformal radiation therapy
Radiation: radiation therapy — 66.6 Gy (1.8 Gy per fraction, 5 days per week) to the prostate bed (IMRT or 3DCRT), starting 8 weeks after start of hormones

SUMMARY:
RATIONALE: Specialized radiation therapy that delivers a high-dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue. Androgens can cause the growth of prostate cancer cells. Antihormone therapy, such as leuprolide, goserelin, flutamide, or bicalutamide, may lessen the amount of androgens made by the body. Drugs used in chemotherapy, such as docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving radiation therapy together with androgen suppression and docetaxel after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This phase II trial is studying how well giving radiation therapy together with androgen suppression and docetaxel works in treating patients with high risk prostate cancer who have undergone radical prostatectomy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess whether the addition of androgen suppression therapy and docetaxel to adjuvant radiotherapy improves freedom from progression.

Secondary

* To assess freedom from local-regional progression, distant metastases, disease-free survival, prostate cancer specific survival, non-prostate cancer specific survival, overall survival, and time to biochemical (PSA) failure.
* To evaluate treatment-related "acute" and "late" toxicity based on Common Toxicity Criteria for Adverse Effects (CTCAE) v3.0.
* To correlate genomic and proteomic biomarkers with the primary and secondary clinical endpoints utilizing archival prostatectomy tissue and pretreatment and prospectively collected serum/plasma.

OUTLINE: This is a multicenter study.

* Androgen suppression therapy: Patients receive a luteinizing hormone-releasing hormone (LHRH) agonist (leuprolide or goserelin) as an injection AND an oral antiandrogen (flutamide 3 times daily or bicalutamide once daily) for up to 6 months.
* Radiotherapy: Beginning 8 weeks after the initiation of androgen suppression therapy, patients undergo 3-dimensional conformal radiotherapy or intensity-modulated radiotherapy once a day 5 days a week for up to approximately 8 weeks.
* Chemotherapy: Beginning 3-6 weeks after the completion of radiotherapy, patients receive docetaxel IV over 1 hour on day 1. Treatment repeats every 21 days for up to 6 courses.

After the completion of study treatment, patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Pathologically proven adenocarcinoma of the prostate gland meeting one of the following criteria:

  * Gleason ≥ 7and post-operative PSA nadir > 0.2 ng/ml with any pathologic tumor (pT) classification
  * Gleason ≥ 8, post-operative PSA nadir ≤ 0.2 ng/ml and ≥ pT3a classification
* Must have undergone radical prostatectomy within the past year
* PSA must be obtained within 6 weeks (42 days) prior to study registration
* No lymph node or distant metastases (N0, M0), based upon the following minimum diagnostic workup:

  * History and physical examination within 8 weeks prior to study registration
  * Bone scan and CT or MRI of the pelvis and no evidence of osseous metastases on bone scan within 16 weeks prior to study registration
* No pelvic lymph nodes > 1.5 cm in greatest dimension on CT scan or MRI of the pelvis within 16 weeks prior to study registration, unless the enlarged lymph node is biopsied and negative

PATIENT CHARACTERISTICS:

* Zubrod performance status 0-1
* Absolute neutrophil count (ANC) ≥ 2,000/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 8.0 g/dL (transfusion or other intervention to achieve hemoglobin ≥ 8.0 g/dL is acceptable)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 2.5 times ULN
* Total bilirubin ≤ 1.2 times ULN
* No other invasive malignancy within the past 3 years except non-melanomatous skin cancer
* No active, severe co-morbidity, including any of the following:

  * Unstable angina and/or congestive heart failure requiring hospitalization within the past 6 months
  * Transmural myocardial infarction within the past 6 months
  * Acute bacterial or fungal infection requiring intravenous antibiotics
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy
  * AIDS

    * HIV testing is not required for study entry
* No prior allergic reaction to the study drug(s)

PRIOR CONCURRENT THERAPY:

* No prior systemic chemotherapy for prostate cancer
* More than 3 years since prior chemotherapy for a different cancer
* No prior androgen deprivation for treatment of prostate cancer

  * Prior use of hormonal agents, such as finasteride or dutasteride, for treatment of benign prostatic hypertrophy is allowed
* No prior radiotherapy to the region of the prostate that would result in overlap of radiotherapy fields

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2008-04 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2018-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Hurwitz, MD, Principal Investigator — Thomas Jefferson University and Hospitals; Oliver Sartor, MD, Study Chair — Dana-Farber Cancer Institute; Ying Xiao, PhD, Study Chair — Bodine Center for Cancer Treatment at Thomas Jefferson University Hospital
Locations (70):
- United States (69):
  - Arizona Oncology Services Foundation, Phoenix, Arizona
  - Auburn Radiation Oncology, Auburn, California
  - Radiation Oncology Centers - Cameron Park, Cameron Park, California
  - Mercy Cancer Center at Mercy San Juan Medical Center, Carmichael, California
  - Radiation Oncology Center - Roseville, Roseville, California
  - Radiological Associates of Sacramento Medical Group, Incorporated, Sacramento, California
  - Mercy General Hospital, Sacramento, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Solano Radiation Oncology Center, Vacaville, California
  - Urology Center of Colorado, Denver, Colorado
  - Poudre Valley Radiation Oncology, Fort Collins, Colorado
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Cancer Institute at St. John's Hospital, Springfield, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Norton Suburban Hospital, Louisville, Kentucky
  - Tulane Cancer Center Office of Clinical Research, Alexandria, Louisiana
  - Mary Bird Perkins Cancer Center - Baton Rouge, Baton Rouge, Louisiana
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Hudner Oncology Center at Saint Anne's Hospital - Fall River, Fall River, Massachusetts
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Regional Cancer Center at Singing River Hospital, Pascagoula, Mississippi
  - Cancer Institute of Cape Girardeau, LLC, Cape Girardeau, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Nevada Cancer Institute, Las Vegas, Nevada
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital Marlton, Marlton, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - University Medical Center at Princeton, Princeton, New Jersey
  - Mission Hospitals - Memorial Campus, Asheville, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Wayne Radiation Oncology, Goldsboro, North Carolina
  - Pardee Memorial Hospital, Hendersonville, North Carolina
  - Cancer Centers of North Carolina - Raleigh, Raleigh, North Carolina
  - Forsyth Regional Cancer Center at Forsyth Medical Center, Winston-Salem, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Barberton Citizens Hospital, Barberton, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Cancer Care Center, Incorporated, Salem, Ohio
  - Precision Radiotherapy at University Pointe, West Chester, Ohio
  - Cancer Treatment Center, Wooster, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Integris Oncology Services, Oklahoma City, Oklahoma
  - St. Luke's Cancer Network at St. Luke's Hospital, Bethlehem, Pennsylvania
  - Delaware County Regional Cancer Center at Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Fox Chase Cancer Center Buckingham, Furlong, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center CCOP Research Base, Philadelphia, Pennsylvania
  - Crozer-Chester Medical Center, Upland, Pennsylvania
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Jon and Karen Huntsman Cancer Center at Intermountain Medical Center, Murray, Utah
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Community Memorial Hospital Cancer Care Center, Menomonee Falls, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
- McGill Cancer Centre at McGill University, Montreal, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Androgen Suppression + RT + Docetaxel: Luteinizing hormone-releasing hormone (LHRH) agonist and oral antiandrogen (flutamide or bicalutamide), radiation therapy (RT), and docetaxel
Period: Overall Study
Arm/Group | Androgen Suppression + RT + Docetaxel
Started | 80
Completed | 74 (Subjects with data available for the primary analysis are considered to have completed the study.)
Not Completed | 6
Not completed — Protocol Violation | 6

BASELINE CHARACTERISTICS:
Population: Eligible and started protocol treatment
Arm/Group | Androgen Suppression + RT + Docetaxel
Number analyzed (Participants) | 74
Age, Continuous [Median (Full Range); unit: years] | 62 [43 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 74

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Free From Progression at 3 Years
Description: Failure was defined as PSA ≥ 0.4 ng/mL after the end of radiation therapy confirmed by a second higher PSA, non-protocol hormones, local-regional progression, distant metastasis, or death, within 3 years after study registration. Freedom from progression (FFP) rate under null hypothesis was 50%; under alternative hypothesis ≥ 70%. Per Fleming's multiple testing procedure with 3 stages, 69 patients (76 allowing for 10% ineligible) were required for 90% power and type I error 0.025. If ≥ 44 of 69 patients had a FFP event, we would reject 50% FFP rate in favor of ≥ 70%. Analysis was out of 74 patients (not 69), so ≥ 44 was revised to ≥ 46.
Time Frame: From registration to 3 years.
Population: All eligible patients who started study treatment
Measure: Number; unit: participants
Arm/Group | Androgen Suppression + RT + Docetaxel
Number analyzed (Participants) | 74
participants | 54

2. Secondary Outcome: Local-regional Progression (3 Year Rate)
Description: Time from registration to date of local progression (failure), death (competing risk), or last follow-up (censored). Three-year failure rate and 95% confidence interval were estimated by the cumulative incidence method.
Time Frame: Analysis occurs after all patients have been on study for at least 3 years. (Patients are followed from registration to death or study termination whichever occurs first.)
Population: All eligible patients who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Androgen Suppression + RT + Docetaxel
Number analyzed (Participants) | 74
percentage of participants | 0 [NA to NA] — A confidence interval cannot be computed when the rate is zero, i.e. when there are zero events.

3. Secondary Outcome: Distant Metastasis (3-year Rate)
Description: Time from registration to date of distant metastasis (failure), death (competing risk), or last follow-up (censored). Three-year failure rate and 95% confidence interval were estimated by the cumulative incidence method.
Time Frame: as for outcome 2
Population: All eligible patients who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Androgen Suppression + RT + Docetaxel
Number analyzed (Participants) | 74
percentage of participants | 6.8 [2.5 to 14]

4. Secondary Outcome: Prostate Cancer Death (3-year Rate)
Description: as for outcome 3
Time Frame: as for outcome 2
Population: All eligible patients who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Androgen Suppression + RT + Docetaxel
Number analyzed (Participants) | 74
percentage of participants | 0 [NA to NA] — A confidence interval cannot be computed when the rate is zero, i.e. when there are zero events.

5. Secondary Outcome: Non-prostate Cancer Death (3-year Rate)
Description: Time from registration to date of death due to other causes (failure), death due to prostate cancer (competing risk), or last follow-up (censored).Three-year failure rate and 95% confidence interval were estimated by the cumulative incidence method.
Time Frame: as for outcome 2
Population: All eligible patients who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Androgen Suppression + RT + Docetaxel
Number analyzed (Participants) | 74
percentage of participants | 1.4 [0.1 to 6.5]

6. Secondary Outcome: Overall Survival (3-year Rate)
Description: Time from registration to date of death (failure) or last follow-up (censored). Three-year rate and 95% confidence interval were estimated by the Kaplan-Meier method.
Time Frame: as for outcome 2
Population: All eligible patients who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Androgen Suppression + RT + Docetaxel
Number analyzed (Participants) | 74
percentage of participants | 98.6 [96 to 100]

7. Secondary Outcome: Time to Biochemical (PSA) Failure (3-year Rate)
Description: Failure is defined as PSA ≥ 0.4 ng/mL confirmed by a second higher PSA or initiation of non-protocol hormones. Death is considered a competing risk. Three-year failure rate and 95% confidence interval were estimated by the cumulative incidence method.
Time Frame: as for outcome 2
Population: All eligible patients who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Androgen Suppression + RT + Docetaxel
Number analyzed (Participants) | 74
percentage of participants | 25.7 [16.3 to 36.1]

8. Secondary Outcome: Number of Patients With "Acute" Adverse Events (Based on CTCAE, v3.0)
Description: The number of patients with at least one grade 3 or higher adverse event (AE) from start of treatment to 90 days after the planned end of treatment (21 days after last docetaxel dose). Adverse events are graded using CTCAE v3.0. Grade refers to the severity of the AE. The CTCAE v3.0 assigns Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild AE, Grade 2 Moderate AE, Grade 3 Severe AE, Grade 4 Life-threatening or disabling AE, Grade 5 Death related to AE.
Time Frame: From start of treatment to 90 days after the planned end of treatment (21 days after last docetaxel dose). Analysis occurs at the time of the primary analysis. (Patients are followed until death or study termination whichever occurs first.
Population: All eligible patients who started study treatment
Measure: Number; unit: participants
Arm/Group | Androgen Suppression + RT + Docetaxel
Number analyzed (Participants) | 74
participants | 57

9. Secondary Outcome: Time to "Late" Grade 3+ Adverse Events (Based on CTCAE, v3.0)
Description: Two-year rate shown (cumulative incidence method). Adverse events are graded using CTCAE v3.0. Time of first late adverse event occurrence of the Grade 3+ adverse event between 91 days and 730 days from the completion of treatment (3 weeks after the last planned docetaxel dose) calculated. Adverse events are graded using CTCAE v3.0. Grade refers to the severity of the AE. The CTCAE v3.0 assigns Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild AE, Grade 2 Moderate AE, Grade 3 Severe AE, Grade 4 Life-threatening or disabling AE, Grade 5 Death related to AE.
Time Frame: From 91 to 730 days after the planned end of treatment (21 days after last docetaxel dose). Analysis occurs at the time of the primary analysis. (Patients are followed from registration to death or study termination whichever occurs first.)
Population: All eligible patients who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Androgen Suppression + RT + Docetaxel
Number analyzed (Participants) | 74
percentage of participants | 8.1 [3.3 to 15.8]

10. Secondary Outcome: Prognostic Value of Genomic and Proteomic Markers for the Primary and Secondary Clinical Endpoints
Time Frame: Analysis can occur at the same time as the primary endpoint if data is available.
Population: The protocol did not provide sufficient detail to meet National Cancer Institute requirements for release of specimens from the NRG tissue bank for the protocol-specified analysis, therefore no assays were performed and no data were collected for this outcome measure. Specimen use will require federal approval and funding separate from this trial.
Arm/Group | Androgen Suppression + RT + Docetaxel
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: Subjects experiencing more than one of a given adverse event are counted only once for that adverse event.
Arm/Group | Androgen Suppression + RT + Docetaxel
Serious Adverse Events (participants affected / at risk) | 20/74
Other Adverse Events (participants affected / at risk) | 73/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Androgen Suppression + RT + Docetaxel (N=74)
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Hemoglobin decreased (Blood and lymphatic system disorders) | 2
Ventricular fibrillation (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Chills (General disorders) | 1
Fatigue (General disorders) | 1
Sinusitis [with normal or Grade 1-2 ANC] (Infections and infestations) | 1
Creatinine increased (Investigations) | 1
Leukopenia (Investigations) | 5
Lymphopenia (Investigations) | 4
Neutrophil count decreased (Investigations) | 7
Dehydration (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Ureteric obstruction (Renal and urinary disorders) | 2
Urinary frequency (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Androgen Suppression + RT + Docetaxel (N=74)
Hemoglobin decreased (Blood and lymphatic system disorders) | 59
Watering eyes (Eye disorders) | 6
Abdominal pain (Gastrointestinal disorders) | 5
Constipation (Gastrointestinal disorders) | 33
Diarrhea (Gastrointestinal disorders) | 51
Dyspepsia (Gastrointestinal disorders) | 10
Fecal incontinence (Gastrointestinal disorders) | 5
Flatulence (Gastrointestinal disorders) | 5
Gastrointestinal disorder (Gastrointestinal disorders) | 9
Hemorrhoids (Gastrointestinal disorders) | 6
Mucositis oral (Gastrointestinal disorders) | 13
Nausea (Gastrointestinal disorders) | 34
Proctitis (Gastrointestinal disorders) | 12
Rectal hemorrhage (Gastrointestinal disorders) | 6
Rectal pain (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 12
Chills (General disorders) | 7
Edema limbs (General disorders) | 35
Fatigue (General disorders) | 70
Fever (General disorders) | 10
General symptom (General disorders) | 5
Localized edema [trunk/genital] (General disorders) | 8
Pain [NOS] (General disorders) | 4
Pain [other] (General disorders) | 11
Dermatitis radiation (Injury, poisoning and procedural complications) | 5
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 6
Alanine aminotransferase increased (Investigations) | 10
Aspartate aminotransferase increased (Investigations) | 11
Creatinine increased (Investigations) | 7
Laboratory test abnormal (Investigations) | 9
Leukopenia (Investigations) | 40
Lymphopenia (Investigations) | 23
Neutrophil count decreased (Investigations) | 44
Platelet count decreased (Investigations) | 16
Weight gain (Investigations) | 12
Weight loss (Investigations) | 5
Anorexia (Metabolism and nutrition disorders) | 15
Dehydration (Metabolism and nutrition disorders) | 7
Hyperglycemia (Metabolism and nutrition disorders) | 39
Hyperkalemia (Metabolism and nutrition disorders) | 5
Hypoalbuminemia (Metabolism and nutrition disorders) | 7
Hypocalcemia (Metabolism and nutrition disorders) | 5
Hypokalemia (Metabolism and nutrition disorders) | 4
Hyponatremia (Metabolism and nutrition disorders) | 14
Arthritis (Musculoskeletal and connective tissue disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 15
Bone pain (Musculoskeletal and connective tissue disorders) | 15
Joint pain (Musculoskeletal and connective tissue disorders) | 25
Muscle weakness (Musculoskeletal and connective tissue disorders) | 8
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 4
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 16
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7
Dizziness (Nervous system disorders) | 14
Headache (Nervous system disorders) | 11
Memory impairment (Nervous system disorders) | 8
Peripheral sensory neuropathy (Nervous system disorders) | 49
Taste alteration (Nervous system disorders) | 29
Agitation (Psychiatric disorders) | 4
Anxiety (Psychiatric disorders) | 8
Depression (Psychiatric disorders) | 12
Insomnia (Psychiatric disorders) | 19
Libido decreased (Psychiatric disorders) | 10
Bladder pain (Renal and urinary disorders) | 4
Cystitis (Renal and urinary disorders) | 13
Urethral pain (Renal and urinary disorders) | 7
Urinary frequency (Renal and urinary disorders) | 56
Urinary incontinence (Renal and urinary disorders) | 42
Urinary retention (Renal and urinary disorders) | 8
Urogenital disorder (Renal and urinary disorders) | 6
Ejaculation disorder (Reproductive system and breast disorders) | 4
Erectile dysfunction (Reproductive system and breast disorders) | 38
Gynecomastia (Reproductive system and breast disorders) | 5
Pelvic pain (Reproductive system and breast disorders) | 6
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 12
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 25
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 6
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 4
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 4
Acne (Skin and subcutaneous tissue disorders) | 6
Alopecia (Skin and subcutaneous tissue disorders) | 47
Dry skin (Skin and subcutaneous tissue disorders) | 13
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 7
Nail disorder (Skin and subcutaneous tissue disorders) | 20
Pruritus (Skin and subcutaneous tissue disorders) | 6
Rash desquamating (Skin and subcutaneous tissue disorders) | 11
Skin disorder (Skin and subcutaneous tissue disorders) | 10
Sweating (Skin and subcutaneous tissue disorders) | 5
Flushing (Vascular disorders) | 4
Hot flashes (Vascular disorders) | 51
Hypertension (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.